CLINICAL TRIAL: NCT04289519
Title: Retrospective Study on Endoscopic Findings of Gastritis in Children Attending GIT Endoscopic Unit of Assiut University Children Hospital (AUCH) (15 Years)
Brief Title: Endoscopic Findings of Gastritis in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, HM Reyad, principle investigator, Assiut University
Other Study IDs: EFOGIC
Record Dates: First submitted 2019-09-23; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Gastritis
MeSH Terms: conditions — Gastritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gastritis defines any (histologically confirmed) inflammation of the gastric mucosa

DETAILED DESCRIPTION:
Gastritis is a very common disease in children. The main presentation of children with gastritis is recurrent abdominal pain and dyspepsia or vomiting. Young children may have hematemesis or melena as presentation. Drug induced or food related gastritis presents usually with acute symptoms but Helicobacter pylori gastritis have mainly recurrent abdominal pain and dyspeptic symptoms. Other presentations include diarrhea, constipation, flatulence, bloating, fatigue, low energy level, weight loss, muscle loss, bad breath etc.

The main causes of gastritis are infections, inflammation and other disorders affect the gastric mucosa in pediatric patients. Helicobacter pylori infection is the most common cause of gastritis in children which is also responsible for the majority of duodenal ulcers.

Acute erosive gastritis is most commonly the result of metabolic stress or drug or corrosive injury.

Other major causes of gastritis include celiac disease, allergic disorders, and Crohn's disease .Medication as NSAIDs, uremia, ischemia, shock, radiation, sepsis, trauma, severe burns and surgery.

Endoscopic pictures in acute gastritis may be in the form of:

* Multiple round-shaped severe erosions with a diameter of several millimeters.
* Mucosal edema, hyperemia.
* Peptic ulcer While in chronic gastritis is variable. Affects the antrum in the beginning and advances to the proximal in time .

ELIGIBILITY:
Inclusion Criteria:

* All children diagnosed as gastritis by upper endoscopy and bio gastric biopsy

Exclusion Criteria:

* • All children underwent upper endoscopy during the study period not diagnosed as gastritis

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All children diagnosed as gastritis by upper endoscopy and bio gastric biopsy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-09-30 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
causes of gastritis in children as shown by upper endoscopy | average 1 year
  * infections
  * inflammation
  * Helicobacter pylori
  * Acute erosive gastritis

REFERENCES:
- [Background] Pasechnikov VD, Chukov SZ, Kotelevets SM, Mostovov AN, Mernova VP, Polyakova MB. Invasive and non-invasive diagnosis of Helicobacter pylori-associated atrophic gastritis: a comparative study. Scand J Gastroenterol. 2005 Mar;40(3):297-301. doi: 10.1080/00365520410010607. PMID 15932170
- [Background] Kusters JG, van Vliet AH, Kuipers EJ. Pathogenesis of Helicobacter pylori infection. Clin Microbiol Rev. 2006 Jul;19(3):449-90. doi: 10.1128/CMR.00054-05. PMID 16847081
- [Background] Gold BD, Colletti RB, Abbott M, Czinn SJ, Elitsur Y, Hassall E, Macarthur C, Snyder J, Sherman PM; North American Society for Pediatric Gastroenterology and Nutrition. Helicobacter pylori infection in children: recommendations for diagnosis and treatment. J Pediatr Gastroenterol Nutr. 2000 Nov;31(5):490-7. doi: 10.1097/00005176-200011000-00007. No abstract available. PMID 11144432
- [Background] Tam YH, Chan KW, To KF, Cheung ST, Mou JW, Pang KK, Wong YS, Sihoe JD, Lee KH. Impact of pediatric Rome III criteria of functional dyspepsia on the diagnostic yield of upper endoscopy and predictors for a positive endoscopic finding. J Pediatr Gastroenterol Nutr. 2011 Apr;52(4):387-91. doi: 10.1097/MPG.0b013e31820e2026. PMID 21415670
- [Background] Glickman JN, Antonioli DA. Gastritis. Gastrointest Endosc Clin N Am. 2001 Oct;11(4):717-40, vii. PMID 11689363
- [Background] Kayacetin S, Guresci S. What is gastritis? What is gastropathy? How is it classified? Turk J Gastroenterol. 2014 Jun;25(3):233-47. doi: 10.5152/tjg.2014.7906. PMID 25141310